CLINICAL TRIAL: NCT05075577
Title: A Phase 1/2 Study of EPI-7386 in Combination with Enzalutamide Compared with Enzalutamide Alone in Subjects with Metastatic Castration-Resistant Prostate Cancer
Brief Title: EPI-7386 in Combination with Enzalutamide Compared with Enzalutamide Alone in Subjects with MCRPC
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was terminated early due to a lack of improved efficacy.
Sponsor: ESSA Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EPI-7386-CS-010
Record Dates: First submitted 2021-09-14; First posted 2021-10-13 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Phase 1 Cohort 1 (Experimental): 600 mg QD EPI-7386 in combination of Enzalutamide120 mg
  Interventions: Drug: EPI-7386 with Enzalutamide
- Phase 1 Cohort 2 (Experimental): 800 mg QD EPI-7386 in combination of Enzalutamide120 mg
  Interventions: Drug: EPI-7386 with Enzalutamide
- Phase 1 Cohort 3 (Experimental): 600 mg BID EPI-7386 in combination of Enzalutamide120 mg
  Interventions: Drug: EPI-7386 with Enzalutamide
- Phase 1 Cohort 4 (Experimental): RP2D mg EPI-7386 in combination of Enzalutamide160 mg
  Interventions: Drug: EPI-7386 with Enzalutamide
- Phase 2 Enzalutamide + EPI-7386 (Randomized 2:1) (Experimental): RP2D mg EPI-7386 in combination of Enzalutamide RP2D mg
  Interventions: Drug: EPI-7386 with Enzalutamide
- Phase 2 Enzalutamide single agent (Active Comparator): Enzalutamide 160 mg
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Enzalutamide — Daily oral dose of enzalutamide
  Arms: Phase 2 Enzalutamide single agent
Drug: EPI-7386 with Enzalutamide — Daily oral dose of EPI-7386 in combination of enzalutamide
  Arms: Phase 1 Cohort 1; Phase 1 Cohort 2; Phase 1 Cohort 3; Phase 1 Cohort 4; Phase 2 Enzalutamide + EPI-7386 (Randomized 2:1)

SUMMARY:
This is a Phase 1/2 study of EPI-7386 orally administered in combination with enzalutamide in subjects with mCRPC.

Phase 1 of the study will be a single-arm dose escalation study of EPI-7386 in combination with a fixed dose of enzalutamide. This portion of the study will primarily evaluate the safety and tolerability of the drug combination and establish the RP2CDs for EPI-7386 and enzalutamide when dosed in combination. In addition, blood sampling will be conducted for PK evaluation to assess the potential DDI between the two drugs.

Once the RP2CD for each drug has been established, Phase 2 of the study will commence. Phase 2 is a two-arm, randomized (2:1), open-label study. Approximately 120 subjects will be randomized 2:1 to:

* Group 1: EPI-7386 at the RP2CD + enzalutamide(depending on the results of the Phase 1) (n=80)
* Group 2: Enzalutamide single agent (n=40) The planned dose of enzalutamide and EPI-7386 for the combination arm will be those determined in the Phase 1 of this study based on safety and exposure data. Subjects may remain on study treatment as long as they are tolerating treatment without disease progression based on RECIST v1.1 and/or PCWG3.

ELIGIBILITY:
Inclusion Criteria:

* Males ≥18 years.
* Histologically, pathologically, or cytologically confirmed prostate adenocarcinoma.
* Evidence of castration-resistant prostate cancer (CRPC).
* Presence of metastatic disease at study entry documented by 1 or more bone lesions on bone scan or by soft tissue disease observed by CT/MRI.
* Naïve to second generation anti-androgens.
* Evidence of progressive disease defined as 1 or more Prostate Cancer Working Group 3 (PCWG3) criteria.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Ongoing ADT with luteinizing hormone-releasing hormone (LHRH) agonist/antagonist therapy or history of bilateral orchiectomy, with castrate level testosterone.
* Serum testosterone ≤1.73 nmol/L (50 ng/dL).
* Subjects receiving bisphosphonates or other approved bone-targeting therapy (e.g., denosumab) must be on a stable dose for at least 28 days prior to the start of study treatment.
* Demonstrate adequate organ function.

Exclusion Criteria:

* Biologic anti-cancer therapy within 28 days prior to the start of study treatment.
* Use of hormonal agents with anti-tumor activity against prostate cancer within 28 days prior to the start of study treatment.
* Use of herbal products or alternative therapies that may decrease PSA levels or that may have hormonal anti-prostate cancer activity within 28 days prior to the start of study treatment or plans to initiate during the study.
* Intervention with any chemotherapy, investigational agents, or other anti-cancer drugs within 28 days of the first dose of study treatment.
* Use of radium-223 dichloride or other radioligand/radiopharmaceutical within 28 days prior to the start of study treatment.
* Received limited-field palliative bone radiotherapy >5 fractions and/or any radiotherapy within 2 weeks prior to the start of study treatment.
* Received a blood transfusion within 28 days of hematologic screening labs.
* Known intra-cerebral disease or brain metastasis unless adequately treated and stable for the last 28 days before signing of informed consent.
* Spinal cord compression.
* Diagnosis of another clinically significant malignancy within the previous 3 years other than curatively treated non-melanomatous skin cancer or superficial urothelial carcinoma and other in situ or non-invasive malignancies.
* Gastrointestinal issues affecting absorption.
* Significant cardiovascular disease.
* Known history of seizure or conditions that may pre-dispose them to seizure, including brain injury with loss of consciousness, transient ischemic attack within the past 12 months, cerebral vascular accident, brain metastases, and brain arteriovenous malformation.
* Concurrent disease or any clinically significant abnormality.
* Known or suspected hypersensitivity to any components of the formulation used for EPI-7386 or enzalutamide.
* Use of strong inhibitors of CYP2C8.
* Use of strong inducers of CYP3A.
* Use of narrow therapeutic index sensitive CYP2C8 or sensitive substrates for CYP3A and CYP2B6.
* Use of granulocyte colony stimulating factor within 7 days prior to screening laboratories.
* Not a candidate for enzalutamide treatment.
* Patients with rare hereditary problems of fructose intolerance.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 77 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-01-14 (Actual)

PRIMARY OUTCOMES:
Phase 1: Incidence of Dose Limiting Toxicities | Baseline to End of Cycle 1 (each cycle is 28 days)
  Characterized by type, frequency, severity (as graded by National Cancer Institute Common Terminology Criteria for AEs [NCI CTCAE version 5.0]), timing in relation to study treatment administration, seriousness, and relationship to study treatment.
Phase 1: Incidence of treatment emergent adverse events | Baseline to 30 days after last dose of study drug
  Characterized by type, frequency, severity, timing, seriousness, and relationship to study treatment.
Phase 1: Incidence of laboratory abnormalities as a measure of safety and tolerability of EPI-7386 | Baseline to 30 days after last dose of study drug
  Characterized by type, frequency, severity, timing, seriousness, and relationship to study treatment.
Phase 1: Changes in ECOG performance status | Baseline to 30 days after last dose of study drug
Phase 2: Proportion of subjects with a prostate-specific antigen decline of >90% (PSA90) at Week 12 | Baseline to Week 12

CONTACTS AND LOCATIONS:
Locations (24):
- United States (13):
  - Arizona Urology, Tucson, Arizona
  - Hematology Oncology Associates of the Treasure Coast, Port Saint Lucie, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Chesapeake Urology Associates, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Washington University Siteman Cancer Center, St Louis, Missouri
  - Urology Cancer Center, Omaha, Nebraska
  - Great Lakes Cancer Center, Buffalo, New York
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - OHSU Knight Cancer Instititue, Portland, Oregon
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - University of Wisconsin, Madison, Wisconsin
- Australia (4):
  - The Canberra Hospital, Garran, Australian Capital Territory
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - St. Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Eastern Health, Box Hill, Victoria
- Canada (7):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Prostate Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Juravinski Cancer Centre, Hamilton, ON L8V 5C2, Hamilton, Ontario
  - Princess Margaret Cancer Center, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec